CLINICAL TRIAL: NCT03108534
Title: A Single Dose, Randomised, Double Blind, Double Dummy, Placebo Controlled, 3-way Crossover Clinical Study, Comparing the Onset of Relief From Methacholine-induced Bronchoconstriction With CHF1535 100/6 µg NEXThaler® Versus CHF1535 100/6 µg pMDI in Asthmatic Patients.
Brief Title: A Study to Evaluate the Onset of Relief From Methacholine-induced Bronchoconstriction With CHF1535 NEXThaler in Asthmatic Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-01535BD1-01; 2016-003672-47 (EudraCT Number)
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHF1535 NEXThaler (Experimental): CHF1535 100/6 NEXThaler (Beclometasone dipropionate 100 µg + formoterol fumarate 6 µg)
  Interventions: Drug: CHF1535 NEXThaler
- CHF1535 pMDI (Active Comparator): CHF1535 100/6 pMDI (Beclometasone dipropionate 100 µg + formoterol fumarate 6 µg)
  Interventions: Drug: CHF1535 pMDI
- Placebo (Placebo Comparator): Double dummy study: placebo is for both CHF1535 pMDI and CHF1535 NEXThaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF1535 NEXThaler — Rescue treatment
  Other Names: Foster NEXThaler
  Arms: CHF1535 NEXThaler
Drug: CHF1535 pMDI — Rescue treatment
  Other Names: Foster
  Arms: CHF1535 pMDI
Drug: Placebo — Rescue treatment
  Arms: Placebo

SUMMARY:
The clinical trial is designed to evaluate the non-inferiority of CHF1535 100/6 µg NEXThaler versus CHF1535 100/6 µg pMDI on the onset of relief from methacholine-induced bronchospasm, in terms of pulmonary function (i.e. change in Forced Expiratory Volume in the 1st second, FEV1, from baseline to 5 min after study drug intake) in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form obtained
* Minimum required Peak Inspiratory Flow (PIF) to activate NEXThaler
* Pre-bronchodilator FEV1 of at least 65%
* Positive response to methacholine challenge test
* Previous treatment with low-medium doses of Inhaled Corticosteroids (ICS) or ICS/Long-acting beta2-agonist (LABA) as per Global Initiative for Asthma (GINA) 2016 guidelines
* For females: non-pregnant, non-lactacting and using highly effective contraceptive methods.

Exclusion Criteria:

* Clinically relevant and uncontrolled concomitant diseases
* Abnormal clinically relevant ECG
* Presence of aortic aneurism
* Uncontrolled hypertension
* Intake of non-permitted concomitant medications
* Participation in another clinical trials in the previous 8 weeks
* Seasonal variation in asthma
* Recent occurrence of asthma exacerbations
* Hypersensitivity to any product used in the trial, including excipients
* Heavy caffeine drinkers
* History of alcohol/drug abuse
* Smokers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 5-min post-dose | 5 min post-dose
  Change in FEV1 from baseline (baseline is the post-diluent value, before methacholine challenge test)

SECONDARY OUTCOMES:
Change in FEV1 other time points | Up to 30 min post-dose
  Change in FEV1 from baseline (baseline is the post-diluent value, before methacholine challenge test)
FEV1 AUC0-10min | From dosing to 10 min post-dose
  FEV1 area under the curve from dosing to 10 min post-dose
Time to recovery in FEV1 | From dosing to 30 min post-dose
  Time to return to 85% of baseline value
Change in Borg scale | Up to 30 min post-dose
  Change in Borg scale from the end of the methacholine challenge test
Time to recovery in Borg scale | Up to 30 min post-dose
  50% decrease from the post-methacholine challenge value

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - University of Dundee, Dundee
  - Hammersmith Medicines Research, London
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-003672-47/results